CLINICAL TRIAL: NCT04722900
Title: PREG-Offspring: Untersuchung Von Kindern Von Teilnehmerinnen Der Deutschen Studie Gestationsdiabetes (PREG-Studie)
Brief Title: PREG - Offspring: Investigation of Children From Mothers With and Without Gestational Diabetes
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: 617/2020BO1
Record Dates: First submitted 2021-01-14; First posted 2021-01-25 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Offspring Exposed to GDM and Control

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-GDM
- GDM
  Interventions: Other: intrauterine exposure to elevated glucose levels

INTERVENTIONS:
Other: intrauterine exposure to elevated glucose levels — intrauterine exposure to elevated glucose levels
  Groups: GDM

SUMMARY:
Gestational diabetes is the most common complication during pregrancy. With a screening between week 24 and 28 of gestation women with gestational diabetes can be identified and treated. Treatment comprises modification of diet and in some cases taking medication. This treatment lowers undesirable events like macrosomia or premature birth. However, unitl gestational diabetes is diagnosed the fetus is exposed to increased intrauterine glucose levels. The long-term effects of a well-managed gestational diabetes on the development of the offspring is still not well understood. Therefore, the PREG - Offspring study investigates several aspects of development in children from healthy and gestational diabetes mothers until adulthood.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent provided by child and parent
* documented oral glucose tolerance test of the mother during pregnancy
* adequate management of gestational diabetes until birth

Exclusion Criteria:

* severe malformation that makes an examination impossible
* existent of coagulation disorder with increased risk of bleeding after blood sampling

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study participants are children from mothers that are enrolled in the PREG study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2036-01-15 (Estimated); Study Completion 2036-09-15 (Estimated)

PRIMARY OUTCOMES:
Body height | Change in body height from birth to age 6, 10, 14 and 17
  Body height is measured with a tape measure in centimeter (cm)

SECONDARY OUTCOMES:
Body weight | Change in body weight from birth to age 6, 10, 14 and 17
  Body weight is measured with a scale in kilogram (kg)
Body fat | Change of body fat from age 6 to age 10, 14 and 17
  Body fat content is measured with bioimpedance anaylsis in percent (%)
Blood pressure | Change of blood pressure from age 6 to age 10, 14 and 17
  Blood pressure is measured with a blood pressure monitor as systolic and diastolic pressure in millimeter mercury column (mm Hg)
Pubertal development scale | Change of pubertal development scale from age 6 to age 10, 14 and 17
  Pubertal development scale is assessed according to Tanner stages
Blood glucose | Change of blood glucose from age 6 to age 10, 14 and 17
  Blood glucose is measured in blood sample in miligram per deciliter (mg/dl)
HbA1C | Change of HbA1C from age 6 to age 10, 14 and 17
  HbA1C is measured in blood sample in percent (%)
Cardiometabolic risk markers | Change of cardiometabolic risk markers from age 6 to 10, 14 and 17
  Cholesterol, Low-density Lipoprotein, High-density Lipoprotein, Triglycerides, Lipoprotein(a) are measured in blood sample in mg/dl
Continuous glucose monitoring | Change of blood glucose from age 6 to age 10, 14 and 17
  24h glucose profiles and postprandial glycemic excursions (AUC) will be measured by flash glucose monitoring
Activity level | Change of activity level from age 6 to 10, 14 and 17
  Activity level is assessed with the MOMO activity questionnaire
Magnetic resonance imaging | Change of magnetic resonance images from age 6 to 10, 14 and 17
  Distribution of whole body fat and visceral and subcutaneous fat confirmed by MR-Imaging and proton magnetic resonance spectroscopy by 3T Whole Body Imager

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Fritsche, Principal Investigator — University Hospital Tübingen
Locations (1):
- University Hospital Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fritsche L, Hummel J, Wagner R, Loffler D, Hartkopf J, Machann J, Hilberath J, Kantartzis K, Jakubowski P, Pauluschke-Frohlich J, Brucker S, Horber S, Haring HU, Roden M, Schurmann A, Solimena M, de Angelis MH, Peter A, Birkenfeld AL, Preissl H, Fritsche A, Heni M. The German Gestational Diabetes Study (PREG), a prospective multicentre cohort study: rationale, methodology and design. BMJ Open. 2022 Feb 15;12(2):e058268. doi: 10.1136/bmjopen-2021-058268. PMID 35168986